CLINICAL TRIAL: NCT03737695
Title: AURORA US: Prospective Biospecimen Repository in Metastatic Breast Cancer
Brief Title: Clinical Information and Biospecimen Collection From Patients With Recurrent or Stage IV Breast Cancer
Status: Suspended | Type: Observational
Why Stopped: enrollment pause
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: AURORA US; NCI-2018-02144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AURORA (Other: Mayo Clinic); 18-001910 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Metastatic Breast Carcinoma; Peritoneal Effusion; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen, clinical info collection): Patients' archival and newly collected tissue and blood samples are collected periodically for genetic testing. Patients also undergo collection of clinical information within 30 days of biopsy procedure and every 4 months.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo biospecimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Medical Chart Review — Undergo clinical information collection
  Other Names: Chart Review

SUMMARY:
This trial collects clinical information and tissue and blood samples from patients with breast cancer that has come back or is stage IV. Collecting clinical information and biospecimen samples to create a registry may help doctors better understand the mechanism of tumor spread and determine why people respond differently to specific cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To create a comprehensive registry that includes patient demographics, clinical and histopathological data, blood samples, and tissue specimens from the primary tumor and metastatic sites of patients with metastatic breast cancer to improve our understanding of the mechanisms of tumor metastasis and therapeutic resistance.

II. To conduct genomic studies of paired primary tumors and distant metastatic sites.

III. To conduct genomic studies of paired distant metastatic sites obtained during the course of an individual's disease.

IV. To conduct genomic studies of cell free deoxyribonucleic acid (DNA), circulating tumor cell (CTC) derived DNA, germline DNA, and immune based markers in the peripheral circulation.

SECONDARY OBJECTIVE:

I. To evaluate the concordance between DNA sequencing results obtained from a clinically available assay and those obtained specifically for research purposes.

OUTLINE:

Patients' archival and newly collected tissue and blood samples are collected periodically for genetic testing. Patients also undergo collection of clinical information within 30 days of biopsy procedure and every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or suspected invasive breast cancer
* Radiographic evidence of distant metastatic disease
* Clinical or radiographic evidence of disease progression OR presenting with de novo stage IV disease
* Available archived tissue from the initial breast primary (formalin fixed paraffin embedded [FFPE] tissue is acceptable; fresh frozen tissue is preferred if available)
* Accessible lesion representative of recurrent or metastatic breast cancer for biopsy

  * Type 1 specimen collection: Patients undergoing a clinically directed tissue biopsy or tissue collection who are willing to have additional specimens taken for research during the same procedure. Sites for tissue acquisition may include the breast, skin/chest wall, lymph node/soft tissue, liver, bone, lung, brain, pleural fluid, and ascites as needed for routine clinical care
  * Type 2 specimen collection: Patients undergoing a tissue biopsy or tissue collection for research purposes only. Sites for tissue acquisition include the breast, skin/chest wall, lymph node/soft tissue, liver, bone, pleural fluid, and ascites. Research directed lung biopsies and brain biopsies are not permitted. Procedures for tissue acquisition are restricted to those performed under local anesthesia or intravenous (IV) conscious sedation; biopsies that require general anesthesia are not permitted in this situation
* Previous cytologic confirmation of malignant pleural effusion or ascites if that is the planned source of fresh specimen collection for study participation
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign an informed consent document

Exclusion Criteria:

* Concurrent disease or condition that in the opinion of the treating oncologist or the provider performing the biopsy procedure renders the patient inappropriate for study participation
* Concurrent serious medical or psychiatric disorder that may interfere with the subject's safety during the biopsy or tissue collection procedure
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* History of a serious or life-threatening allergic reaction to local anesthetics (e.g., lidocaine, xylocaine) used during a biopsy procedure
* Pregnancy (due to the risk of conscious sedation or anesthesia to mother and fetus)
* Any condition or laboratory finding that in the opinion of the treating oncologist or the provider performing the biopsy procedure would make participation in this protocol hazardous for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent and/or metastatic breast cancer of all tumor subtypes
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Comprehensive biorepository creation | Up to 2 years
  Will create a comprehensive biorepository that includes blood, archival tissue, fresh tissue, and linked molecular and clinical data from patients with recurrent and/or metastatic breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Karthik V. Giridhar, M.D., Principal Investigator — Mayo Clinic
Locations (14):
- United States (14):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - FHCC South Lake Union, Seattle, Washington

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials